CLINICAL TRIAL: NCT05031806
Title: A Single-Center, Randomized, Double Masked, Vehicle Controlled Clinical Study to Assess the Safety and Efficacy of iNexin™ Eye Drops Compared to Vehicle in Subjects With Dry Eye Disease
Brief Title: Evaluation of the Safety, Tolerability and Efficacy of iNexin™ for the Treatment of the Signs and Symptoms Associated With Dry Eye Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xequel Bio, Inc. (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-OCLR-01b; CDMRP-VR190131 (Other Grant/Funding Number: DOD)
Record Dates: First submitted 2021-08-17; First posted 2021-09-02 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — TRAF3IP2 protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- iNexin™ (0.08% aCT1) (Experimental): 36 eligible subjects will be randomized to Vehicle or one of three concentrations of iNexin™ to be administered bilaterally BID for 15 days (from Visit 2 to the evening of Visit 4). Subjects will be randomized 2:1 for each active concentration to Vehicle. During a 7-day study run-in period prior to randomization, all subjects will receive Vehicle eye drops (Vehicle) bilaterally BID (from Visit 1 to the evening before Visit 2).
  Interventions: Drug: iNexin™ (0.08% aCT1)
- iNexin™ (0.4% aCT1) (Experimental): 36 eligible subjects will be randomized to Vehicle or one of three concentrations of iNexin™ to be administered bilaterally BID for 15 days (from Visit 2 to the evening of Visit 4). Subjects will be randomized 2:1 for each active concentration to Vehicle. During a 7-day study run-in period prior to randomization, all subjects will receive Vehicle eye drops (Vehicle) bilaterally BID (from Visit 1 to the evening before Visit 2).
  Interventions: Drug: iNexin™ (0.4% aCT1)
- iNexin™ (2.0% aCT1) (Experimental): 36 eligible subjects will be randomized to Vehicle or one of three concentrations of iNexin™ to be administered bilaterally BID for 15 days (from Visit 2 to the evening of Visit 4). Subjects will be randomized 2:1 for each active concentration to Vehicle. During a 7-day study run-in period prior to randomization, all subjects will receive Vehicle eye drops (Vehicle) bilaterally BID (from Visit 1 to the evening before Visit 2).
  Interventions: Drug: iNexin™ (2.0% aCT1)
- Vehicle (eye drop formulation without aCT1) (Placebo Comparator): 36 eligible subjects will be randomized to Vehicle or one of three concentrations of iNexin™ to be administered bilaterally BID for 15 days (from Visit 2 to the evening of Visit 4). Subjects will be randomized 2:1 for each active concentration to Vehicle. During a 7-day study run-in period prior to randomization, all subjects will receive Vehicle eye drops (Vehicle) bilaterally BID (from Visit 1 to the evening before Visit 2).
  Interventions: Drug: Vehicle (eye drop formulation without aCT1)

INTERVENTIONS:
Drug: iNexin™ (0.08% aCT1) — 36 eligible subjects will be randomized to Vehicle or one of three concentrations of iNexin™ to be administered bilaterally BID for 15 days (from Visit 2 to the evening of Visit 4). Subjects will be randomized 2:1 for each active concentration to Vehicle.randomized 7:3 for each active concentration to Vehicle.
  Arms: iNexin™ (0.08% aCT1)
Drug: iNexin™ (0.4% aCT1) — 36 eligible subjects will be randomized to Vehicle or one of three concentrations of iNexin™ to be administered bilaterally BID for 15 days (from Visit 2 to the evening of Visit 4). Subjects will be randomized 2:1 for each active concentration to Vehicle.
  Arms: iNexin™ (0.4% aCT1)
Drug: iNexin™ (2.0% aCT1) — 36 eligible subjects will be randomized to Vehicle or one of three concentrations of iNexin™ to be administered bilaterally BID for 15 days (from Visit 2 to the evening of Visit 4). Subjects will be randomized 2:1 for each active concentration to Vehicle.
  Arms: iNexin™ (2.0% aCT1)
Drug: Vehicle (eye drop formulation without aCT1) — 36 eligible subjects will be randomized to Vehicle or one of three concentrations of iNexin™ to be administered bilaterally BID for 15 days (from Visit 2 to the evening of Visit 4). Subjects will be randomized 2:1 for each active concentration to Vehicle.
  During a 7-day study run-in period prior to randomization, all subjects will receive Vehicle eye drops (Vehicle) bilaterally BID (from Visit 1 to the evening before Visit 2).
  Arms: Vehicle (eye drop formulation without aCT1)

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of iNexin™ The secondary objective is to compare the efficacy of iNexin™ to Vehicle for the treatment of the signs and symptoms associated with dry eye disease.

DETAILED DESCRIPTION:
The clinical hypothesis for this study is that iNexin™ demonstrates safety and tolerability in subjects with DED and can be evaluated for further safety and efficacy measures compared to vehicle. This is a Phase 1b single-center, randomized, double masked, vehicle controlled clinical study to assess the safety and exploratory efficacy of iNexin™ compared to vehicle in subjects with Dry Eye Disease. A total of 36 subjects, at least 18 years of age, with a subject-reported history of DED in both eyes and meeting all other study eligibility criteria will be randomized to receive treatment with iNexin™ or vehicle.

An individual subject's participation time is expected to be approximately 24 days. 36 eligible subjects will be randomized in a 2:1 allocation for each of three concentrations of iNexin™ to Vehicle, to be administered bilaterally BID for 15 days (from Visit 2 to the evening of Visit 4). There will also be a 1-day post-final dose follow-up visit (Visit 5).

During a 7-day study run-in period prior to randomization (from Visit 1 to the evening before Visit 2), all subjects will receive Vehicle eye drops (Vehicle) bilaterally at the same dosing frequency as iNexin™ (BID).

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following requirements to be eligible for enrollment into the study.

1. Be at least 18 years of age;
2. Provide written informed consent;
3. Have a self-reported history of dry eye for at least 6 months prior to Visit 1;
4. Have a history of use or desire to use eye drops for dry eye symptoms for at least 6 months prior to Visit 1;
5. Report a score of ≥ 2 according to a 0-5 point scale in at least one symptom of the Ora Calibra Ocular Discomfort & 4-Symptom Questionnaire pre-CAE at Visits 1 and 2;
6. Have a conjunctival redness score of ≥ 1 according to a 0-4 point scale in at least one eye at Visits 1 and 2;
7. Have a tear film break-up time (TFBUT) >1 and < 7 seconds in at least one eye pre-CAE at Visit 1 and 2;
8. Have an unanesthetized Schirmer's Test score of ≤ 10 mm and ≥ 1 mm in at least one eye pre-CAE at Visits 1 and 2;
9. Have a corneal fluorescein staining sum of ≥ 6 according to a 0-4 point scale (sum of inferior, superior, and central) in at least one eye pre-CAE at Visits 1 and 2;
10. Have a central corneal fluorescein staining score of ≥ 1 according to a 0-4 point in at least one eye pre-CAE at Visits 1 and 2;
11. Have a total lissamine green conjunctival score of ≥ 2, based on the sum of the temporal and nasal regions of the conjunctiva according to a 0-4 point scale in at least one eye pre-CAE at Visits 1 and 2;
12. Demonstrate a response to the CAE at Visits 1 and 2 as defined by:

    1. Having at least a ≥ 1 point increase in fluorescein staining in the inferior region in at least one eye following CAE exposure; and
    2. Reporting an Ocular Discomfort score ≥ 3 at 2 or more consecutive time points in at least one eye during CAE exposure (if a subject has an Ocular Discomfort rating of 3 at time = 0 for an eye, s/he must report an Ocular Discomfort rating of 4 for two consecutive measurements for that eye).
13. Have at least one eye (the same eye) satisfy all criteria for 6, 7, 8, 9, 10, 11, and 12 above.

Exclusion Criteria:

Subjects may not participate in the study if any of the following criteria are met:

1. Unable or unwilling to follow instructions, including participation in all study assessments and visits;
2. Have active blepharitis, meibomian gland dysfunction (MGD) or lid margin inflammation that required any topical or systemic antibiotics or topical steroids or other prescription medical treatment or treatment with hypochlorous acid wipes within the last 3 months prior to Visit 1 or will require such treatment during the trial.

   Any other therapy such as lid scrubs, lid wipes, warm compresses have to be stable within the last 3 months prior to Visit 1 and the subject should be willing to continue those therapies through the trial
3. Have active ocular allergies that require therapeutic treatment, and/or in the opinion of the Investigator may interfere with study parameters;
4. Be diagnosed with an ongoing ocular infection (bacterial, viral, or fungal), or active ocular inflammation at Visit 1;
5. Have a significant ocular lesion that the investigator feels might affect ocular surface staining score;
6. Have worn contact lenses within 14 days of Visit 1 or anticipate using contact lenses during the study;
7. Have previously had laser-assisted in situ keratomileusis (LASIK) or any other Laser refractive surgery within the last 12 months or any other ocular surgeries within the last 6 months;
8. Have any planned ocular and/or lid surgeries over the study period;
9. Current smoker (includes tobacco, marijuana, or vaping) or has smoked within 6 months of Visit 1;
10. Has dry eye secondary to known systemic diseases or comorbidities:

    1. Previous diagnosis of graft versus host disease or cicatrizing conjunctivitis (e.g., Steven-Johnson Syndrome, mucous membrane pemphigoid, trachoma, trauma);
    2. Anatomical or neurological lid closure problems (e.g., Bell's palsy, cicatricial ectropion, Alzheimer's disease, Parkinson's disease);
11. Has dry eye secondary to other ocular surface diseases or ocular surgery:

    1. Ocular rosacea, blepharitis, demodex infestation, atopic keratoconjunctivitis, etc.;
    2. Any history of surgery for glaucoma (e.g., trabeculectomy, tube shunt);
    3. Cataract, eyelid surgery, or retinal surgery (in operating room) within 6 months prior to enrollment;
    4. Any in-office dry eye procedures (e.g., Intense Pulsed Light [IPL], LipiFlow , nasolacrimal duct probing) within 90 days prior to enrollment;
12. Has a history of corneal dystrophy that in the opinion of the investigator is significantly affecting the ocular surface (e.g., significant anterior basement membrane dystrophy, Fuch's dystrophy with significant corneal edema and bullae, neurotrophic keratoconjunctivitis or corneal/conjunctival scarring including herpes simplex virus [HSV] or varicella zoster virus [VZV] keratitis);
13. Has any physical or mental condition interfering with the successful participation in this study;
14. Has had any past head and neck radiation treatment;
15. Be using or anticipate using temporary punctal plugs;
16. Be using or anticipate using permanent punctal plugs during the study that have not been stable within 3 months of Visit 1;
17. Have had punctal occlusion (other than permanent punctal plugs) within 6 months of Visit 1;
18. Have corrected visual acuity greater than or equal to logMAR+0.7 as assessed by Early Treatment of Diabetic Retinopathy Study (ETDRS) scale in either eye at Visit 1
19. Have an uncontrolled systemic disease;
20. Be a woman who is pregnant, nursing or planning a pregnancy;
21. Be unwilling to submit a urine pregnancy test at Visit 1 and Visit 5 (or early termination visit) if a woman of childbearing potential (WOCBP). Non-childbearing potential is defined as a woman who is permanently sterilized (e.g. has had a hysterectomy or tubal ligation), or is post-menopausal (without menses for 12 consecutive months);
22. Be a woman of childbearing potential (WOCBP) who does not have a negative pregnancy test at Screening or who does not agree to use an acceptable means of birth control; acceptable methods of contraception include: hormonal - oral, implantable, injectable, or transdermal contraceptives; mechanical - spermicide in conjunction with a barrier such as a diaphragm or condom; IUD; surgical sterilization of partner; For non-sexually active females, abstinence may be regarded as an adequate method of birth control; however, if the subject becomes sexually active during the study, she must agree to use adequate birth control as defined above for the remainder of the study. Male subjects must abstain from sex with WOCBP or use an adequate method of contraception (as described above) from the time of informed consent through the end of the study;
23. Have a known allergy and/or sensitivity to the test article or its components;
24. Have a condition or be in a situation which the Investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study;
25. Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 30 days of Visit 1;
26. Have used any of the following treatments in the period indicated before Visit 1 or anticipate their use at any time during the study: Day of Visit 1 1. All topical ophthalmic preparations (e.g., over-the counter-solutions, artificial tears, gels, scrubs, ointments) 7 days prior to Visit 1 2. Antihistamines (including topical ophthalmic antihistamines) 3. Medications for glaucoma 30 days prior to Visit 1 4. Topical ophthalmic non-steroidal anti-inflammatories 5. Topical ophthalmic corticosteroids 6. Topical ophthalmic autologous serum 7. Topical ophthalmic antibiotics 8. Mast cell stabilizers (Zaditor and Alamast ) 9. Oral aspirin or aspirin-containing products except in the case that it was taken on a stable daily dosing regimen for at least 30 days prior to Visit 1 and is expected to be taken on the same regimen throughout the study period 10. Any other medication known to cause ocular drying (e.g., anticholinergics, diuretics, antidepressants, beta blockers) except in the case that it was taken on a stable daily dosing regimen for at least 30 days prior to Visit 1 and is expected to be taken on the same regimen throughout the study period 12 weeks prior to Visit 1 11. Restasis 12. Xiidra 13. CEQUA™ 14. Eysuvis™ 15. LipiFlow or other similar meibomian gland dysfunction (MGD) therapy 16. TrueTear 17. Corticosteroids (e.g., systemic steroids including intravenous, intramuscular, intraarticular, and oral steroids; facial topical steroids; dermatological steroids with high potency or large treatment areas); 18. Tetracyclines (tetracycline, doxycycline, minocycline, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the safety of iNexin™ | Through study completion, an average of 24 days
  Assessed using: Visual Acuity (VA) (ETDRS), Slit-lamp biomicroscopy, Adverse Event Query, Dilated Fundoscopy Interocular Pressure
Evaluation of the tolerability of iNexin™ | Through study completion, an average of 24 days
  Assessed using: Ora Calibra Drop Comfort Assessments

SECONDARY OUTCOMES:
Comparison of the efficacy of iNexin™ to Vehicle for the treatment of the signs and symptoms associated with dry eye disease | Through study completion, an average of 24 days
  Efficacy measures: Corneal fluorescein staining using the Ora Calibra Corneal and Conjunctival Staining Scale, Conjunctival lissamine green staining using the Ora Calibra Corneal and Conjunctival Staining Scale, Visual Analogue Scale (VAS) for symptoms, Tear film break-up time (TFBUT), Ora Calibra Conjunctival Redness, Unanesthetized Schirmer's Test, Ora Calibra Ocular Discomfort Scale, Ora Calibra Ocular Discomfort & 4- Symptom Questionnaire; OSDI

CONTACTS AND LOCATIONS:
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No